CLINICAL TRIAL: NCT06962332
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of Zanzalintinib in Participants With Moderate Hepatic Impairment
Brief Title: Pharmacokinetics (PK) and Safety of Zanzalintinib in Participants With Moderate Hepatic Impairment (HI)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL092-008
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Impairment; Moderate Hepatic Impairment
Keywords: Zanzalintinib; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate HI (Experimental): Participants with moderate HI will receive a single oral dose of zanzalintinib tablet on Day 1.
  Interventions: Drug: Zanzalintinib
- Matched Healthy Control (Active Comparator): Matched healthy control participants will receive a single oral dose of zanzalintinib tablet on Day 1.
  Interventions: Drug: Zanzalintinib

INTERVENTIONS:
Drug: Zanzalintinib — Administered as specified in the treatment arm.
  Other Names: XL092

SUMMARY:
The primary purpose of this study is to evaluate the plasma PK of zanzalintinib following a single dose in participants with moderate liver dysfunction compared to matched healthy participants with normal liver function.

ELIGIBILITY:
Key Inclusion Criteria:

* All Participants:

  * No clinically significant medical history (aside from the HI for participants in the HI group only), physical examination findings, or vital signs, as deemed by the investigator.
  * A continuous non-smoker or moderate smoker who smokes ≤ 10 cigarettes, ≤ 2 cigars, or ≤2 pipes per day and agree to limit smoking during the confinement period to ≤ 4 cigarettes or ≤1 cigar or pipe per day. Participant must agree to maintain the same smoking status (smoker or non-smoker) from screening and until after the last PK sample collection.
  * Has not donated blood within 30 days of dosing or plasma within 7 days of dosing and must agree to refrain from blood donation until at least 30 days following dosing.
* Participants with Moderate HI Only:

  * Adequate bone marrow function, at the screening and dosing visit.
  * Is classified as having moderate HI by the Child-Pugh classification system (Class B, score of 7 to 9, inclusive) and has a total bilirubin value within the range of > 1.5* upper limit of normal (ULN) and ≤ 3* ULN at the screening and dosing visit.
  * Has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency at the screening visit with features of cirrhosis due to any etiology.
* Healthy Control Participants Only:

  * Age must be within ± 10 years of the mean age of participants with moderate HI. The sex ratio (male/female ratio), and smoking status ratio (smokers/non-smokers ratio) must be the same to the sex and smoking status ratio of participants with moderate HI.

Key Exclusion Criteria:

* All Participants:

  * • History of any medical or surgical conditions that would potentially alter absorption, distribution, metabolism, and/or excretion of orally administered drugs.
  * Has or is at risk for major cardiac events or dysfunction.
* Participants with Moderate HI Only:

  * History of liver or other solid organ transplant.
  * Fluctuating or rapidly deteriorating hepatic function (the definition of the change of more than 1 Child-Pugh point) within 30 days prior to Day 1, in the opinion of the investigator and Sponsor.
  * Symptoms or history of Grade 3 or worse degree of encephalopathy within 3 months of dosing.
  * Clinical evidence of severe ascites at the screening visit or at check in.
* Healthy Control Participants Only:

  * History or presence of alcohol or drug abuse within the past 2 years prior to dosing.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Time t Corresponding to the Last Quantifiable Concentration (AUC0-t) of Zanzalintinib | Predose up to 7 days postdose
Maximum Observed Plasma Drug Concentration (Cmax) of Zanzalintinib | Predose up to 7 days postdose
Time to Cmax (Tmax) of Zanzalintinib | Predose up to 7 days postdose

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (2):
- United States (2):
  - Exelixis Clinical Site #1, Orlando, Florida
  - Exelixis Clinical Site #2, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No